CLINICAL TRIAL: NCT06670690
Title: Comparison Between Atenolol , Propnalol and Ivabradine as a Premedication for Bloodless Field Anesthesia in Lumbar Spine Surgery ,a Prospective Randomized Controlled Trial
Brief Title: Comparison Between Atenolol,Propnalol and Ivabradine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, Principal investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9/2023ANET 13
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Intraoperative Bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Atenolol; Propranolol; Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atenolol Group (Active Comparator): patients will be premedicated with atenolol (50mg)
  Interventions: Drug: Atenolol 50 MG
- propranolol Group (Active Comparator): patients will be premedicated with propranolol (10mg)
  Interventions: Drug: Propranolol Pill
- Ivabradine Group (Active Comparator): patients will be premedicated with Ivabradine (5mg)
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Atenolol 50 MG — patients will be premedicated with atenolol (50mg)
  Arms: Atenolol Group
Drug: Propranolol Pill — patients will be premedicated with propranolol (10mg)
  Arms: propranolol Group
Drug: Ivabradine — patients will be premedicated with Ivabradine (5mg)
  Arms: Ivabradine Group

SUMMARY:
The aim of this work is to compare atenolol, propranolol, and ivabradine as a premedication to achieve bloodless field anesthesia primarily controlling heart rate in lumbar spine surgery.

DETAILED DESCRIPTION:
This study will investigate the effect of atenolol, propranolol, and ivabradine as oral premedication in adult patients undergoing LUMBAR SPINE SURGERY to achieve bloodless field anesthesia.

AIM OF THE WORK

* The primary aim of this work is to compare atenolol, propranolol, and ivabradine as a premedication to achieve bloodless field anesthesia primarily controlling heart rate in lumbar spine surgery.
* The secondary aims are to assess field visibility and measure the amount of blood loss in patients, and surgeon satisfaction and also to asses if there are any associated undesirable side effects of atenolol, propranolol, or Ivabradine will appear.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II,

  * aged from 18 to 50 years old
  * scheduled for elective lumber spine surgeries will be included in this study.

Exclusion Criteria:

* Hypertension.
* Hepatic or renal disease.
* Diabetes Mellitus.
* Pregnancy.
* Coagulation disorders.
* Anemia (Hb < 10 g/dL).
* Ischemic heart disease
* Drug or alcohol abuse.
* Allergy to any of atenolol, propranolol, and ivabradine.
* History of beta-blockers, calcium channel blockers, Tricyclic antidepressants, anticoagulant or clonidine intake.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Perioperative Heamodynamic Effect of the drugs | every 5 minutes for 15 minutes and then every 10 minutes till end of surgery, then every 15 minutes for 1hour in the recovery room
  Heart rate

SECONDARY OUTCOMES:
Blood loss & surgical field visibility score | Intraoperative time
  quality scale proposed by Fromm and Boezaart
Anesthetic consumption | Intraoperative time
  Propofol, opioid, and isoflurane consumption
Incidence of complication | Intraoperative time
  The patient will be examined for bradycardia, or tachycardia hypo or hypertension, shivering, respiratory depression, dizziness, visual disturbance, nausea, and vomiting
The need for blood transfusion | Intraoperative time
  The need for blood transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Shepien El Kom, Menoufia Government, Egypt

IPD SHARING:
Plan to Share IPD: No